CLINICAL TRIAL: NCT06647732
Title: Zanubrutinib Plus Rituximab as Front-line Treatment for Mucosa-associated Lymphoid Tissue Lymphoma (MALT): a Single-arm, Open-label, Multicenter, Phase II Study（ZAMA）
Brief Title: Zanubrutinib Plus Rituximab as Front-line Treatment for Mucosa-associated Lymphoid Tissue Lymphoma (MALT)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Gansu Cancer Hospital (Other); Fifth Affiliated Hospital of Guangzhou Medical University (Other); Beijing Tongren Hospital (Other); Tongji Medical College of Huazhong University of Science & Technology (Unknown); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Shenzhen People's Hospital (Other)
Responsible Party: Principal Investigator, Qingqing Cai, chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2024-594-01
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-10

CONDITIONS: Mucosa-associated Lymphoid Tissue Lymphoma (MALT)
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — zanubrutinib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zanubrutinib in combination with Rituximab (Experimental): Eligible patients will receive:
  1. Rituximab: 375 mg/m², administered once a week during Cycle 1 (C1), and on Day 1 (D1) of Cycles 2-6 (C2-C6).
  2. Zanubrutinib: 160 mg, administered twice daily from Day 1 to Day 28 (D1-D28). Each cycle lasts 28 days. After 6 cycles of treatment, patients who achieve complete remission (CR) will end treatment and enter observation follow-up, while patients with partial remission (PR) or stable disease (SD) will receive an additional 2 cycles.
  Interventions: Drug: Zanubrutinib; Drug: Rituximab

INTERVENTIONS:
Drug: Zanubrutinib — 160 mg, administered twice daily from Day 1 to Day 28 (D1-D28)
Drug: Rituximab — 375 mg/m², administered once a week during Cycle 1 (C1), and on Day 1 (D1) of Cycles 2-6 (C2-C6)

SUMMARY:
This is a prospective, single-arm, multicenter, phase II clinical trial to evaluate the efficacy and safety of Zanubrutinib in combination with Rituximab as a first-line treatment for patients with mucosa-associated lymphoid tissue (MALT) extranodal marginal zone lymphoma.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and safety of Zanubrutinib in combination with Rituximab as a first-line treatment for patients with mucosa-associated lymphoid tissue (MALT) extranodal marginal zone lymphoma.

Treatrment:

1. Rituximab: 375 mg/m², administered once a week in Cycle 1 (C1) and on Day 1 (D1) of Cycles 2-6 (C2-C6).
2. Zanubrutinib: 160 mg, administered twice daily from Day 1 to Day 28 (D1-D28). Each cycle lasts 28 days. After 6 cycles of treatment, patients who achieve complete remission (CR) will end treatment and enter observation follow-up. Patients with partial remission (PR) or stable disease (SD) will receive 2 additional cycles.

The primary study endpoint is the complete remission rate of Zanubrutinib in combination with Rituximab in the treatment of newly diagnosed mucosa-associated lymphoid tissue (MALT) extranodal marginal zone lymphoma.

ELIGIBILITY:
Key inclusion Criteria:

1. Mucosa-associated lymphoid tissue (MALT) extranodal marginal zone lymphoma confirmed by histopathology.
2. Newly diagnosed with Ann Arbor stage III-IV or relapsed MALT after local treatment .
3. No prior systemic anti-lymphoma therapy (except for H. pylori eradication therapy in H. pylori-positive gastric MALT patients).
4. No histopathological transformation to high-grade lymphoma.
5. At least one measurable lesion according to the Lugano 2014 criteria.

7. Age ≥ 18 years, with no gender restrictions. 7. An ECOG performance status score of 0-2. 8. An expected survival time of more than 12 months. 9. Adequate bone marrow, cardiac, pulmonary, liver, and kidney function. 10. Willing to participate in the clinical study; fully informed and aware of the study, having signed the informed consent form; willing and able to comply with all study procedures.

Key exclusion Criteria:

1. Patients with a history of stroke, intracranial hemorrhage, or warfarin use within the past 6 months.
2. Patients with central nervous system involvement.
3. Patients who have undergone allogeneic hematopoietic stem cell transplantation in the past.
4. Patients who have previously used BTK inhibitors or received CD20 monoclonal antibody therapy.

5, Patients with active infections, except for tumor-related B-symptom fever. 6. Patients with a concurrent history of other malignancies, except for cured cervical carcinoma in situ or basal cell carcinoma of the skin.

7. Patients receiving potent cytochrome P450 inhibitors. 8. Patients with severe cardiovascular diseases, such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or a history of myocardial infarction within the past 12 months.

9. Patients, as judged by the investigator, who have significant organ dysfunction or uncontrollable comorbidities that pose a safety risk, or who have absorption and metabolism issues with Zanubrutinib.

10. Pregnant or breastfeeding women and women of childbearing age unwilling to use contraception.

11. Patients who have received anti-tumor therapy within 4 weeks prior to enrollment.

12. Patients with active chronic hepatitis B or active hepatitis C. 13. Patients who have received systemic corticosteroid treatment or other immunosuppressive therapy within 14 days prior to the start of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Complete Response(CR) | Up to 8 cycles (each cycle is 28 days)
  Defined as the proportion of patients who achieve complete remission as the best response

SECONDARY OUTCOMES:
Objective response rate(ORR) | Up to 8 cycles (each cycle is 28 days)
  The proportion of patients who achieve complete remission (CR) or partial remission (PR) as the best response.
Progression-free survival(PFS) | From the date of enrollment until the date of the first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  To investigate the preliminary anti-tumor efficacy
Event-free survival(EFS) | The proportion of patients without disease progression, treatment discontinuation, or death for any reason since enrollment, assessed up to 24 months
  To investigate the preliminary anti-tumor efficacy
Overall survival(OS) | From the date of enrollment until the date of death from ant cause, assessed up to 24 months
  To investigate the preliminary anti-tumor efficacy
Duration of Response(DOR) | The time from the patient's first efficacy assessment achieving CR or PR until disease progression, assessed up to 24 months
  To investigate the preliminary anti-tumor efficacy
Time to Response(TTR) | The time from the start of patient enrollment in the trial to the first efficacy assessment achieving CR or PR, assessed up tp 24 months
  To investigate the preliminary anti-tumor efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Universitiy Cancer Center, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided